CLINICAL TRIAL: NCT01782066
Title: Dose Finding and Reactogenicity of Reduced-dose Intradermal Administration of Two Quadrivalent Meningococcal Conjugate Vaccines (Menveo® and Nimenrix®) in Healthy Adults (MENID-1).
Brief Title: Dose-finding and Safety of 2 Intradermal MEN-ACYW135-conjugate Vaccines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, L.G. Visser, MD, PhD, Associate professor of Internal Medicine, Senior Consultant Infectious Diseases, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MENID-1; 2012-003085-41 (EudraCT Number)
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Meningococcal Disease
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Menveo, dose escalating (Experimental)
  Interventions: Biological: MEN-ACYW135 reduced-dose intradermal administration
- Nimenrix, dose escalating (Experimental)
  Interventions: Biological: MEN-ACYW135 reduced-dose intradermal administration

INTERVENTIONS:
Biological: MEN-ACYW135 reduced-dose intradermal administration — Modified traditional dose escalation rule (TER) in an adaptive design. The study will be performed in duplicate, with 2 vaccines.
  Other Names: Menveo; Nimenrix

SUMMARY:
Invasive meningococcal disease is a worldwide problem with serious repercussions for those affected. Vaccination is recognized as the best way to combat it. The cost of vaccination is prohibitive in many low-resource settings at home and abroad. By harnessing the special immunologic properties of the skin, a dose reduction may be achieved by intradermal administration of the vaccine. The cost savings associated with dose reduction will increase availability of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

Meningococcal C naive subjects are required to fulfill all of the following criteria:

* Age ≥ 30 years
* Good health according to the investigator
* Willingness and ability to adhere to the study regimen
* Able to give informed consent

Meningococcal C experienced subjects are required to fulfill all of the following criteria:

* Age ≥ 18 years
* Good health according to the investigator
* Willingness and ability to adhere to the study regimen
* Able to give informed consent

Exclusion Criteria:

Meningococcal C naïve subjects should not have:

* Known previous invasive meningococcal infection
* Known or suspected previous vaccination against meningococcal disease
* Known or suspected allergy against any of the vaccine components
* Close contact in the last 60 days with a person known to be Neisseria positive
* History of unusual or severe reactions to any previous vaccination
* Family history of Guillain-Barré Syndrome
* Known or suspected immune deficiency, either congenital or acquired
* Administration of plasma or blood products less than three months prior to inclusion in the study
* Pregnancy (breastfeeding is allowed)
* Fertile female not conforming to prescribed contraceptive use (await first menstruation after vaccination before getting pregnant)
* Any infectious disease
* Bleeding disorders or use of anticoagulants
* Participation as a subject in another trial in the last 3 months

Meningococcal C experienced subjects should not have:

* Known or suspected allergy against any of the vaccine components
* Known previous vaccination with a quadrivalent meningococcal vaccine (either conjugate or polysaccharide)
* Close contact in the last 60 days with a person known to be Neisseria positive
* History of unusual or severe reactions to any previous vaccination
* Family history of Guillain-Barré Syndrome
* Known or suspected immune deficiency, either congenital or acquired
* Administration of plasma or blood products less than three months prior to inclusion in the study
* Pregnancy (breastfeeding is allowed)
* Fertile female not conforming to prescribed contraceptive use (await first menstruation after vaccination before getting pregnant)
* Any infectious disease
* Bleeding disorders or use of anticoagulants
* Participation as a subject in another trial in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate against meningococcal serogroups ACYW135 (anti-meningococcal antibody titre at baseline and 28 days after vaccination) | 28 days

SECONDARY OUTCOMES:
Local and systemic adverse events (subject log and investigator inspection). | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Leo Visser, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

REFERENCES:
- [Derived] Jonker EFF, van Ravenhorst MB, Berbers GAM, Visser LG. Safety and immunogenicity of fractional dose intradermal injection of two quadrivalent conjugated meningococcal vaccines. Vaccine. 2018 Jun 18;36(26):3727-3732. doi: 10.1016/j.vaccine.2018.05.064. Epub 2018 May 16. PMID 29778515